CLINICAL TRIAL: NCT00304759
Title: A Randomized Trial of a Shorter Radiation Fractionation Schedule for the Treatment of Localized Prostate Cancer
Brief Title: PROFIT - Prostate Fractionated Irradiation Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Trans Tasman Radiation Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCOG-2005-PROFIT; CIHR grant MCT-78776; ISRCTN43853433
Record Dates: First submitted 2006-03-17; First posted 2006-03-20 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2016-12

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; localized prostate cancer; intermediate risk; prostate specific antigen; PSA; radiation fractionation; shorter schedule; quality of life
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 6000 cGy / 20 fractions in 4 weeks
  Interventions: Procedure: 6000 cGy/20 fractions in 4 weeks
- 2 (Active Comparator): 7800 cGy / 39 fractions in 8 weeks
  Interventions: Procedure: 7800 cGy/39 fractions in 8 weeks

INTERVENTIONS:
Procedure: 7800 cGy/39 fractions in 8 weeks — see above
  Other Names: standard
  Arms: 2
Procedure: 6000 cGy/20 fractions in 4 weeks — see above
  Other Names: short fractionation schedule
  Arms: 1

SUMMARY:
This trial is designed to determine whether an 8-week course of escalated dose conformal radiation can be compressed safely, and with similar efficacy into a 4-week course.

DETAILED DESCRIPTION:
In this trial, men with intermediate risk prostate cancer will be randomized to a shorter course of radiotherapy (6000cGy in 20 fractions over 4 weeks-hypofractionated) or treatment with a conventional fractionation course (7800cGy in 39 fractions over 8 weeks-standard). Three-dimensional conformal radiation treatment techniques, including intensity modulated radiotherapy will be used for both hypofractionated and standard treatments to avoid normal tissue exposure to radiation and minimize the risk of acute and late treatment related toxicity. The primary outcome measure is biochemical (PSA) failure defined by the ASTRO consensus criteria. Secondary outcomes include biochemical-clinical failure (BCF), mortality from cancer, toxicity and health-related quality of life. It is planned to recruit 1204 patients to the study. If the safety and efficacy of the shorter course are demonstrated, then its adoption would reduce the social, emotional and economic burden of treatment for patients and their families.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of carcinoma of the prostate within 6 months of entry without evidence of metastatic disease to the lymph nodes, bone or lung;
2. Intermediate risk prostate cancer (that is, T1-2a, Gleason score <6, PSA 10.1-20.0 ng/ml; T2b-c Gleason <6, PSA ≤ 20.0 ng/ml; T1-2, Gleason 7, PSA ≤ 20.0 ng/ml).

Exclusion Criteria:

1. Histologic diagnosis of carcinoma of the prostate more than six months prior to study entry;
2. Previous therapy for carcinoma of the prostate other than biopsy or transurethral resection;
3. Patients previously on more than 12 weeks of hormone therapy for treatment of their prostate cancer;
4. Any other active malignancy (untreated, progressive or recurrent), except for non-melanoma skin cancer. Any inactive malignancy diagnosed within 5 years of entry, except for non-melanoma skin cancer;
5. Treatment plan cannot meet dose constraints for the hypofractionation arm of the trial;
6. Previous pelvic radiotherapy;
7. Inflammatory bowel disease.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1204 (Estimated)
Dates: Start 2006-05; Primary Completion 2017-07-15 (Actual); Study Completion 2017-07-15 (Actual)

PRIMARY OUTCOMES:
Biochemical (PSA) Failure | five years

SECONDARY OUTCOMES:
Biochemical-Clinical Failure | five years
Prostate Cancer Specific Mortality | five years
Toxicity | five years
Quality of Life | five years

CONTACTS AND LOCATIONS:
Overall Officials: Charles Catton, MD, Principal Investigator — Princess Margaret Hospital, Canada; Himu Lukka, MD, Principal Investigator — Juravinski Cancer Centre; Mark Levine, MD, Study Director — Ontario Clinical Oncology Group (OCOG); Jim Julian, MMATH, Principal Investigator — McMaster University - Department of Oncology
Locations (25):
- Australia (9):
  - Liverpool Hospital & Campbelltown Hospital, Liverpool, New South Wales
  - Calvary Mater Newcastle Hospital, Newcastle, New South Wales
  - Northern Sydney Cancer Centre, Royal North Shore Hospital, St Leonards, New South Wales
  - Westmead Cancer Care Centre, Wentworthville, New South Wales
  - Wollongong Hospital / Illawarra Cancer Care Centre, Wollongong, New South Wales
  - Toowoomba Cancer Research Centre, Toowoomba, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Ballarat Austin Radiation Oncology Centre (BAROC), Ballarat, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Canada (15):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Centre, London, Ontario
  - The Credit Valley Hospital - Carlo Fidani Peel Regional Cancer Centre, Mississauga, Ontario
  - Stronach Regional Cancer Centre, Southlake Regional Health Centre, Newmarket, Ontario
  - R.S. McLaughlin Durham Regional Cancer Centre, Oshawa, Ontario
  - Odette Sunnybrook Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - CHUM - Hôpital Notre-Dame, Montreal, Quebec
  - Montréal General Hospital, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- Centre René Gauducheau, Nantes, Saint Herblain, France

REFERENCES:
- [Background] Martin J, Frantzis J, Chung P, Langah I, Crain M, Cornes D, Plank A, Finch T, Jones M, Khoo E, Catton C. Prostate radiotherapy clinical trial quality assurance: how real should real time review be? (A TROG-OCOG Intergroup Project). Radiother Oncol. 2013 Jun;107(3):333-8. doi: 10.1016/j.radonc.2013.05.015. Epub 2013 Jun 8. PMID 23751377
- [Derived] Sanmamed N, Dayes I, Catton C, Liu A, Supiot S, Lukka H, Bauman G, Liu Z, Bahary JP, Ahmed S, Cheung P, Parliament M, Sia M, Tsakiridis T, Siva S, Corbett T, Tang C, Craig T, Martin J, Chung P. Patient-reported Quality of Life in PROFIT, a Phase 3 Randomized Clinical Trial Evaluating Moderately Hypofractionated Radiotherapy for Intermediate-risk Prostate Cancer. Eur Urol Oncol. 2025 May 6:S2588-9311(25)00095-1. doi: 10.1016/j.euo.2025.03.017. Online ahead of print. PMID 40335398